CLINICAL TRIAL: NCT04585451
Title: Expanded Development of a Medical Device Utilizing an EEG-Based Algorithm for the Objective Quantification of Pain
Status: Completed | Type: Observational
Sponsor: PainQx, Inc (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: PQXNIH2; 5R44DA046964-03 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Chronic Pain Patients
  Interventions: Diagnostic Test: ALGOS System
- Healthy Controls
  Interventions: Diagnostic Test: ALGOS System

INTERVENTIONS:
Diagnostic Test: ALGOS System — A Quantitative Electroencephalography (QEEG) based pain biomarker assessment that scales with patient reported Numeric Rating Scale (NRS)

SUMMARY:
PainQx is conducting a study to collect electroencephalography (EEG) data from 250 people with chronic pain and 50 healthy controls in order to develop algorithms that will objectively assess the level of pain a person is experiencing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female chronic pain patients
* Patients between the ages of 18-85 years
* Patients exhibiting the presence of symptoms in excess of 3 months duration
* Patients suffering from neuropathic (e.g., lower back pain), osteoarthritis, or muscular skeletal pain
* Patients with evidence of pathology related to the painful condition on which diagnosis was made (e.g., results of imaging or diagnostic pain code)

Patients with NRS pain scores across the full range (1-10) at the time of testing Inclusion Criteria, Normal (no-pain) Group

o Subjects will be included with no history of pain with a duration of greater than 3 months, and no report of pain at the time of testing (or within 3 months of testing)

Exclusion Criteria:

* Patients with medically diagnosed psychotic illness
* Patients with medically diagnosed drug or alcohol dependence in the past 12 months
* Patients with a medical history of head injury with loss of consciousness and amnesia (within the last 2 years)
* Patients with skull abnormalities that preclude the proper placement of the electrodes for the EEG data acquisition
* Patients who have a spinal cord stimulator, or other implantable devices
* Patients for whom the source of pain at the time of the evaluation is associated with: neurological disorders (multiple sclerosis, Parkinson, dementia), diabetes, migraines, or those with reflex / sympathetic dystrophy disorder/complex regional pain syndrome, fibromyalgia, or visceral pain

Note: This does not exclude patients who suffer from these disorders if the current source of pain is not due to the disorder. For example, patients with diabetes are NOT excluded, but patients whose pain at the time of the evaluation is a result of diabetic neuropathy are excluded. Similarly, patients with a history of migraines but for whom a migraine is not the current source of pain at the time of the evaluation are NOT excluded.

* Patients with cancer
* Patients on workers compensation or disability
* Patient on anticonvulsant medication
* Patients who have a history of seizures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two hundred fifty (250) male and female pain patients with symptoms in excess of 3 months duration (per the IASP definition of Chronic Pain) between the ages of 18-85 years will be enrolled in this phase of the study. Fifty (50) healthy normal subjects between the ages of 18-85 years will also be enrolled. The normal subjects are added to assure that the study spans the entire pain scale including those with an NRS of 0.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Koppes, Principal Investigator — PainQx, Inc
Locations (5):
- United States (5):
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - Comprehensive Spine and Pain Center of New York, New Hyde Park, New York
  - Pain Management at Comprehensive Pain and Wellness Center, New York, New York
  - Comprehensive Spine and Pain Center of New York, New York, New York
  - Comprehensive Spine & Pain Center of New York, Valley Stream, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Pain Patients | Healthy Controls
Started | 280 | 54
Completed | 254 | 54
Not Completed | 26 | 0
Not completed — Withdrawal by Subject | 26 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chronic Pain Patients: Chronic pain patients who meet the IASP definition of chronic pain for a musculoskeletal pain disorder.
- Healthy Controls: Healthy control participants with no diagnosis of chronic pain nor other various neurological conditions
- Total: Total of all reporting groups
Arm/Group | Chronic Pain Patients | Healthy Controls | Total
Number analyzed (Participants) | 280 | 54 | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 179 | 51 | 230
  >=65 years | 101 | 3 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 34 | 179
  Male | 135 | 20 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 10 | 15 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 80 | 11 | 91
  White | 123 | 26 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 65 | 2 | 67
Region of Enrollment [Number; unit: participants]
  United States | 280 | 54 | 334

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Classification Versus Patient Self Report of Pain vs no Pain State
Description: This measure is the performance of the classification of pain vs no pain compared to the patient self-report in the form of Numerical Rating Scale (NRS). The primary outcome measure is Area Under the Curve (AUC), derived from the Receiver Operating Characteristic (ROC) curve, a standard metric of performance for binary classifiers. AUC is a numeric quantity ranging from 0 to 1, where the value of 1 indicates perfect separation, while 0.5 represents zero separation. AUC represents a fundamental expression of classifier separation performance without the complexity of threshold selection. (NRS 0 vs 1-10)
Time Frame: Self-reported pain using average of NRS value at the start and end of EEG collection, and classification based on 15 minutes of EEG collection.
Population: Analysis was carried out using both arms combined: a control arm (negative class), and a pain arm (positive class). The reason for combining both arms is to assess the classifier's ability to differentiate the two classes and all outcome measures represent the performance of classification.
Measure: Number; unit: probability
Groups:
- Study Participants: All participants in study, chronic pain patients and controls
Arm/Group | Study Participants
Number analyzed (Participants) | 308
probability | .70

2. Primary Outcome: Sensitivity of Classification Versus Patient Self Report of Pain vs no Pain State
Description: Sensitivity, or true positive rate is the probability of a positive result in the true chronic pain patients. This measure is calculated by dividing true positives by the summation of true positives and false negatives. (NRS 0 vs 1-10)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: probability
Arm/Group | Study Participants
Number analyzed (Participants) | 308
probability | .783

3. Primary Outcome: Specificity of Classification Versus Patient Self Report of Pain vs no Pain State
Description: Specificity, or true negative rate is the probability of a negative result in the true healthy control patients. This measure is calculated by dividing true negatives by the summation of true negatives and false positives. (NRS 0 vs 1-10)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: probability
Arm/Group | Study Participants
Number analyzed (Participants) | 308
probability | .607

4. Secondary Outcome: Area Under the Curve of Classification Versus Patient Self Report of no/Mild Pain vs Moderate/Severe Pain State
Description: This measure is the performance of the classification of No/Mild vs Moderate/Severe pain compared to the patient self-report in the form of Numerical Rating Scale (NRS). The outcome measure is Area Under the Curve (AUC), derived from the Receiver Operating Characteristic (ROC) curve, a standard metric of performance for binary classifiers. AUC is a numeric quantity ranging from 0 to 1, where the value of 1 indicates perfect separation (the classifier is correct on every subject), while 0.5 represents zero separation (no better than guessing). AUC represents a fundamental expression of classifier separation performance without the complexity of threshold selection. (NRS 0-3.5 vs 4-10)
Time Frame: as for outcome 1
Population: Analysis was carried out using both arms combined: No/Mild vs Moderate/Severe pain. The reason for combining both arms is to assess the classifier's ability to differentiate the two classes and all outcome measures represent the performance of classification.
Measure: Number; unit: probability
Arm/Group | Study Participants
Number analyzed (Participants) | 308
probability | .694

5. Secondary Outcome: Area Under the Curve of Classification Versus Patient Self Report of no, Mild, or Moderate Pain vs Severe Pain State
Description: This measure is the performance of the classification of No/Mild/Moderate vs Severe pain compared to the patient self-report in the form of Numerical Rating Scale (NRS). The outcome measure is Area Under the Curve (AUC), derived from the Receiver Operating Characteristic (ROC) curve, a standard metric of performance for binary classifiers. AUC is a numeric quantity ranging from 0 to 1, where the value of 1 indicates perfect separation (the classifier is correct on every subject), while 0.5 represents zero separation (no better than guessing). AUC represents a fundamental expression of classifier separation performance without the complexity of threshold selection. (NRS 0-6.5 vs 7-10)
Time Frame: as for outcome 1
Population: Analysis was carried out using both arms combined: No/Mild/Moderate vs Severe pain. The reason for combining both arms is to assess the classifier's ability to differentiate the two classes and all outcome measures represent the performance of classification.
Measure: Number; unit: probability
Arm/Group | Study Participants
Number analyzed (Participants) | 308
probability | .669

ADVERSE EVENTS:
Time Frame: 1 year post recruitment
Description: Observational study without risk of mortality as result of study
Arm/Group | Chronic Pain Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/280 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/280 | 0/54
Other Adverse Events (participants affected / at risk) | 0/280 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04585451/Prot_000.pdf